CLINICAL TRIAL: NCT07128602
Title: Determining the Effects of Non-invasive Brain Stimulation to Improve Quadriceps Muscle Function After ACL Reconstruction.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcadia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ryan Zarzycki, Associate Professor, Arcadia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Arcadia University; 1R15HD118518-01 (NIH)
Record Dates: First submitted 2025-08-14; First posted 2025-08-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation; Quadriceps Muscle Function
Keywords: acl; acl reconstruction; corticospinal excitability; non-invasive brain stimulation

STUDY DESIGN:
Intervention Model Description: Triple-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Active Comparator): This group will receive 20 minutes of active anodal tDCS
  Interventions: Device: active transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): This group will receive sham anodal tDCS. The tDCS unit will be active for the first 30 seconds and the last 30 seconds only.
  Interventions: Device: sham transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: active transcranial direct current stimulation (tDCS) — 20 minutes of anodal tDCS over the primary motor cortex contralateral to the participants surgical limb during a quadriceps torque matching task
  Arms: Active tDCS
Device: sham transcranial direct current stimulation (tDCS) — Participants receive sham tDCS in which the device only delivers current during the first and last 30 seconds while participants perform a quadriceps torque matching task
  Arms: Sham tDCS

SUMMARY:
After knee surgery for a torn ACL, many women struggle with weak thigh muscles for years, partly due to reduced brain signals to these muscles. Our research tests a new approach to improve recovery by using low-level brain stimulation to boost these signals. The investigators will study 42 women, aged 18-35, who had ACL surgery. They'll be split into two groups: one receiving real brain stimulation and another getting a placebo, both during thigh-strengthening exercises. Over six sessions, the investigators measure thigh muscle strength, speed, and steadiness, plus two brain signal measures, using special equipment. The investigators will also check if stronger brain signals lead to better muscle performance, especially in women. Our goal is to show that this new method strengthens thigh muscles better than standard rehab, helping women recover better after surgery. If successful, this could improve physical therapy for women recovering from ACL surgery, making daily activities and return to sport easier.

DETAILED DESCRIPTION:
Quadricep muscle impairments persist for years after anterior cruciate ligament reconstruction (ACLR). Recent evidence suggests that lower neural drive, (i.e., lower corticospinal excitably (CSE)), is associated with pronounced quadriceps muscle performance deficits, which are more severe in females recovering from ACLR than in males. Current postoperative rehabilitation protocols do not target lower neural drive, which can be achieved through non-invasive brain stimulation. Thus, the long-term goal of this research is to improve the effectiveness of ACLR rehabilitation. The objective of this project is to determine if neural drive is the critical missing link in ACLR rehabilitation. To meet this objective, the investigators will administer anodal transcranial direct current stimulation (tDCS), a type of non-invasive brain stimulation known to increase CSE. The investigators will then assess whether it improves three measures of quadriceps muscle performance (in Aim 1) and two measures of CSE (in Aim 2). In Aim 3, the investigators will determine the relationship between observed changes in quadriceps muscle performance and CSE in female participants recovering from ACLR. These aims will be achieved using a randomized, triple-blinded clinical trial with 42 female individuals after ACLR between the ages of 18 and 35 years. All participants will receive six sessions of active or sham anodal tDCS while they perform isolated quadriceps exercises on an isokinetic dynamometer. The two measures of CSE (i.e. active motor threshold and the slope of transcranial magnetic stimulation (TMS) induced recruitment curves) will be determined using surface electromyography on the vastus medialis and TMS. Three measures of quadriceps performance (i.e. peak torque normalized to body weight, rate of torque development (RTD) from 0-100ms and 100-200ms, and torque steadiness) will be determined following standard isometric muscle testing on an isokinetic dynamometer with the hips flexed to 90° and the knees flexed to 60°.

ELIGIBILITY:
Inclusion Criteria:

- females 2-6 months after ACL reconstruction

Exclusion Criteria:

* multiple ligament reconstruction
* osteochondral procedures
* any previous lower extremity surgery
* previous ACL injury
* Metal or implants in the head or neck
* history of neurological disease
* seizures
* severe migraines
* concussion within the last 6 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-04 (Estimated)

PRIMARY OUTCOMES:
Peak quadriceps muscle torque | Pre and post intervention
  Peak torque during a 5 second maximal voluntary isometric contraction
Corticospinal excitability (Slope) | Pre and post intervention
  Slope of a TMS induced stimulus-response curve

SECONDARY OUTCOMES:
Rate of Torque Development (RTD) | Pre and post intervention
  RTD of a maximal voluntary isometric contraction from onset to 100ms (RTD100) and from 100 to 200ms (RTD200) will be used.
Corticospinal excitability (Active Motor Threshold) | Pre and post intervention
  The lowest stimulator intensity needed to produce consistent MEPs >/= 100 microvolts while the participant maintains an isometric contraction at 5% of their MVIC

CONTACTS AND LOCATIONS:
Locations (1):
- Ryan Zarzycki, Glenside, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will submit all primary and secondary outcome data to DASH at the completion of all data collections and prior to any publications. Demographic data including age, sex, and activity level will also be uploaded to DASH.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available no later than time of an associated publication or end of the performance period, whichever comes first. Data will be available indefinitely, based on the repository policy.
Access Criteria: Anyone with access to DASH will be able to examine the data including researchers interested in study replication.

REFERENCES:
- [Background] Leung A, Kantak S, Hammoud S, Abraham R, Zarzycki R. Sex differences in corticospinal excitability and quadriceps performance after anterior cruciate ligament reconstruction. J Orthop Res. 2024 Apr;42(4):769-776. doi: 10.1002/jor.25725. Epub 2023 Nov 27. PMID 37938095
- [Background] Zarzycki R, Leung A, Abraham R, Hammoud S, Perrone M, Kantak S. Determining the safety, feasibility, and effects of anodal transcranial direct current stimulation on corticospinal excitability and quadriceps performance after anterior cruciate ligament reconstruction: a randomized crossover design. Ann Jt. 2025 Jan 21;10:3. doi: 10.21037/aoj-24-15. eCollection 2025. PMID 39981427